CLINICAL TRIAL: NCT04029597
Title: Examining the Use of a Remote Patient Monitoring System in Pediatric Obesity
Brief Title: Remote Patient Monitoring in Pediatric Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0083
Record Dates: First submitted 2019-07-12; First posted 2019-07-23 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity | interventions — Remote Patient Monitoring

STUDY DESIGN:
Intervention Model Description: open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Remote Patient Monitoring (Experimental): Families participating in the study will receive standard medical care as well as the Remote Patient Monitoring System.
  Interventions: Behavioral: Remote Patient Monitoring

INTERVENTIONS:
Behavioral: Remote Patient Monitoring — Families participating in the study will receive standard medical care as well as the RPMS. The RPMS was developed in collaboration with the University of Mississippi Medical Center (UMMC) Center of Telehealth. Patients enrolled in this open trial of the RPMS will interact with the RPMS system on a daily basis and with UMMC's Center for Telehealth nurse care coordinators and research and clinical staff on an as needed basis. The RPMS will provide patients with include an electronic tablet (i.e., iPad) and the ability to receive data from the patient's weight scale and pedometer. Patients will be asked to wear the pedometer daily to track engagement in physical activity and weigh themselves weekly to track weight during the 3 month period. Educational information specific to pediatric obesity and healthy eating and engagement in physical activity will be presented daily through brief presentations and video clips.

SUMMARY:
The goal of this study is to examine the feasibility and efficacy of a remote patient monitoring system for children who are obese.

DETAILED DESCRIPTION:
Pediatric obesity is a critical public health issue, as almost one-third of U.S. youth are overweight and about 17% are obese. Childhood obesity is associated with numerous co-morbid health conditions and psychological maladjustment and medical costs associated with treatment are staggering. Mississippi has the highest rates of overweight and obesity in youth 2 to 19 years of age (over 44%). There is an important need for research to focus on treatments that prevent the development of chronic medical conditions in children at risk, specifically those who are obese and receiving specialty care to reduce morbidity and mortality.

Standard care in multidisciplinary pediatric obesity clinics results in improved weight status in some youth. Remote patient monitoring system (RPMS) technology facilitates patient observations outside of clinical settings; thus, increasing access to medical information and medical care, and reducing health care costs. Use of RPMS in adult chronic illness populations has resulted in improved health outcomes but the implementation and examination of RPMS in pediatric populations has been limited. Mississippi is a rural state, which limits access to medical care in pediatric specialty clinics. The implementation of novel, technology-based strategies is needed to supplement current care to prevent long-term morbidity and reduce health care costs. There is a significant need to examine whether a RPMS is feasible and efficacious in a pilot sample of youth who are obese, which will provide support for larger external grant applications further evaluating the RPMS, as well as to inform clinical care in Mississippi and across the country.

Purpose The main objective of this study is to pilot test a RPMS designed to provide supplemental health care to youth who are obese and receiving specialty medical care in a multidisciplinary pediatric obesity clinic. An open trial of the RPMS will enroll 50 children 8 to 17 years of age who are obese and attending a multidisciplinary pediatric obesity clinic and their parents. During the study, participating youth will receive standard care in the clinic and the RPMS, which will consist of an iPad, weight scale, and pedometer, to use for a 3-month period. The initial feasibility of providing the RPMS in combination with standard clinical care will be evaluated, as well as patient satisfaction. The initial efficacy of the RPMS at improving health related outcomes will also be examined. Families will complete pre-treatment (baseline), post-treatment (Month 3), and three month follow-up (Month 6) assessments consisting of weight status, dietary intake, physical activity, health-related quality of life, self-efficacy, and the home-food environment. Health outcomes (e.g., blood pressure, hemoglobin A1c, glucose) routinely assessed through standard medical care in the clinic will be obtained from child medical charts.

Specific Aims

The goals of the current study are to:

* Assess initial feasibility and satisfaction of implementing a RPMS with children attending a multidisciplinary pediatric obesity clinic.

  o Hypothesis: High feasibility is expected with use of the RPMS and satisfaction rates over 75%.
* Examine initial efficacy of using the RPMS for three months in youth attending a multidisciplinary pediatric obesity clinic (N = 50).

  * Hypothesis 1.1: After the 3-month period and at follow-up, children will exhibit improved weight status, blood pressure, glucose, A1c, dietary intake, physical activity, health-related quality of life, and self-efficacy compared to pre-treatment.
  * Hypothesis 1.2: Parents will report improved child health-related quality of life and home-food environment after the 3-month treatment and follow-up period compared to pre-treatment.

ELIGIBILITY:
Inclusion Criteria:

* child 8 to 17 years of age attending an outpatient pediatric obesity clinic visit,
* child weight status in the obese range (body mass index equal to or above the 95th percentile for age and gender)
* parent and child are fluent in English.

Exclusion Criteria:

* child or parent history of cognitive impairment (developmental delay or intellectual disability) by parent report that would impact ability to understand and complete questionnaires or interact with the RPMS
* child medical condition reported by parents that may prohibit wearing of the actigraph device (e.g., pacemaker).

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 94 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of using the RPMS | Post-Treatment (3 months)
  percent of queries answered and percent of health data collected from the RPMS via the weight scale and pedometer
Satisfaction with using the RPMS | Post-Treatment (3 months)
  ratings from child and parent satisfaction questionnaire developed for use in the study

SECONDARY OUTCOMES:
Weight Status | Post-Treatment (3 months) and Follow-up (6 months)
  BMI z-score change
Blood Pressure | Post-Treatment (3 months) and Follow-up (6 months)
  Systolic and Diastolic clinic assessed
Glucose | Post-Treatment (3 months) and Follow-up (6 months)
  clinic assessed
A1c | Post-Treatment (3 months) and Follow-up (6 months)
  clinic assessed
Dietary Intake | Post-Treatment (3 months) and Follow-up (6 months)
  24 hour dietary recall
Physical Activity | Post-Treatment (3 months) and Follow-up (6 months)
  actigraph assessed
Health-related Quality of Life | Post-Treatment (3 months) and Follow-up (6 months)
  child and parent report from PedsQL
Self-efficacy | Post-Treatment (3 months) and Follow-up (6 months)
  Child Report - combined summed total scores from Child Dietary Self-Efficacy Scale and Self-Efficacy for Physical Activity Scale, total scores range from 20-60, higher scores indicate higher self efficacy
Home food environment | Post-Treatment (3 months) and Follow-up (6 months)
  Parent-report

CONTACTS AND LOCATIONS:
Overall Officials: Crystal Lim, PhD, Principal Investigator — UMMC
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

REFERENCES:
- [Derived] Lim C, Rutledge L, Sandridge S, King K, Jefferson D, Tucker T. Design, Implementation, and Examination of a Remote Patient Monitoring System for Pediatric Obesity: Protocol for an Open Trial Pilot Study. JMIR Res Protoc. 2021 Jul 28;10(7):e29858. doi: 10.2196/29858. PMID 34319245